CLINICAL TRIAL: NCT04078165
Title: Suspended Personal Protection System Versus Conventional Protection (Aka Zero-Gravity vs Shield and Apron)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maarit Venermo, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/09/01
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Radiation Exposure
Keywords: radiation protection; EVAR; endovascular surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero-Gravity (Experimental): In this group, the operator uses the Zero-Gravity protection system
  Interventions: Device: Zero-Gravity
- Conventional (Active Comparator): In this group, the operator uses conventional radiation protection
  Interventions: Device: Conventional radiation protection

INTERVENTIONS:
Device: Zero-Gravity — Free-floating, suspended personal radiation protection
  Arms: Zero-Gravity
Device: Conventional radiation protection — Standard lead shields and aprons
  Arms: Conventional

SUMMARY:
This trial investigates operator radiation doses when performing standardized procedures using two different means of radiation protection, namely conventional lead shield and apron versus suspended protection system (Zero-Gravity, ZG). The performed procedure is standard endovascular aortic repair (EVAR). The hypothesis is that ZG offers superior protection for the operator.

DETAILED DESCRIPTION:
Endovascular aneurysm repair (EVAR) is less invasive than open surgery, yet the procedure causes sustained radiation exposure to the operator and has a potential risk of radiation-induced skin damage and later malignancy. The deterministic (threshold limited) adverse effects of radiation have been known since the invention of the X-ray in 1895, but the stochastic (non-threshold limited) adverse effects are not so apparent and thus need constant refinement. Diligent usage of radiation protection and abidance to ALARA (As Low As Reasonably Achievable) principles minimizes cumulative radiation exposure.

The lens of the human eye is very sensitive to radiation and cataract formation has been reported among medical interventional practitioners. Previous research into differences between conventional protection (apron and shields) and suspended personal protection (Zero Gravity, ZG) claims superior protection, especially to the lens, while using a suspended personal protection system. Ancillary lead glasses may be needed to fully protect the eyes. In other studies randomization of methods was deemed irrelevant due to expected dramatic differences between conventional and suspended protection systems. In addition standardization of procedures was lacking, because of cohort matching difficulties. The methods of measuring scattered radiation varies among previous studies and we have found the evaluation methods flawed.

The aim of this research is to evaluate the total radiation exposure to the interventionalist and assistant during infrarenal abdominal aortic aneurysm stent-grafting, while using either conventional protection (lead apron and shield) or a suspended personal protection system (Zero-Gravity, ZG). The ZG system consists of a lead shield that is suspended from the ceiling or a separate hanger that permits freedom of motion of the operator, and with no weight supported by the operator.

The total radiation doses have seen considerate reduction already in Helsinki, Finland and lower doses may influence the efficacy of the ZG system. Improper usage of the ZG protection gear as a whole can lead to inefficient protection.

The operator's subjective ergonomic feel and experience will be evaluated with a postoperative questionnaire.

The patients will be randomized into two groups: one where the operator will be using conventional protection (shield and apron) and one where the operator will be using the ZG system. The data will be collected during a four month period, which includes approximately 50 standardized EVAR operations.

Dosimeters will be used to collect the data during the procedures and are placed in various anatomical regions (eye, chest, leg, stomach, control outside protection). The exposure dosage to the eye is measured with EYE-D (Eye lens TLD dosimeter) and other measurements are done using DIS-1 dosimeters. Other data collected includes total fluoroscopy duration, total dose area product (DAP), entrance skin air KERMA (ESAK), and body mass index.

The anonymity and rights of participants will be protected. The health of patients is of uttermost importance and there is no difference in care received.

The planning and design has started since May 2019. Data collection will commence after dosimeter testing in September 2019 and last until December 2019. After data analysis the results will be disseminated in Spring 2020. Literature review will take place parallel to the research.

ELIGIBILITY:
Inclusion Criteria:

* all patients eligible for standard EVAR at Helsinki University Hospital

Exclusion Criteria:

* any additional interventions such as embolization, recanalization, screw fixation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Radiation exposure | During operations
  Radiation dosages in multiple dosimeters on operator

SECONDARY OUTCOMES:
Fluoroscopy duration | During operation
  Duration of fluoroscopy in seconds
Fluoroscopy dose area product (DAP) | During operation
  Patient radiation exposure
Entrance skin air KERMA | During operation
  Patient radiation exposure

CONTACTS AND LOCATIONS:
Overall Officials: Maarit Venermo, MD, PhD, Study Director — University of Helsinki
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serna Santos J, Kaasalainen T, Laukontaus S, Bjorkman P, Heinola I, Laine M, Vikatmaa P, Pekkarinen A, Venermo M, Aho P. The Effect of a Suspended Radiation Protection System on Occupational Radiation Doses During Infrarenal EVAR Procedures: A Randomised Controlled Study. Eur J Vasc Endovasc Surg. 2024 Mar;67(3):435-443. doi: 10.1016/j.ejvs.2023.08.039. Epub 2023 Aug 22. PMID 37611731